CLINICAL TRIAL: NCT04987762
Title: An Open-Label, Multicenter, Multiple-Dose, Safety and Tolerability Study of Adhansia XR® Extended-Release Capsules in Children 4 to 12 Years of Age
Brief Title: Safety and Tolerability Study of Adhansia XR® Extended-Release Capsules in Children
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: due to administrative reasons not related to efficacy or safety.
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADA4004
Record Dates: First submitted 2021-07-15; First posted 2021-08-03 (Actual); Results first posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-07

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: ADHD; methylphenidate; Adhansia XR; Pediatric
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adhansia XR (Experimental): Adhansia XR capsules taken orally once daily in the morning
  Interventions: Drug: Adhansia XR

INTERVENTIONS:
Drug: Adhansia XR — Methylphenidate extended-release capsules taken once daily (12.5 mg, 25 mg, 35 mg, 45 mg, 55 mg, and 70 mg)

SUMMARY:
The purpose of this study is to assess the long-term safety of Adhansia XR in children and to characterize the pharmacokinetics (PK) in 4 to 5 year-olds.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥4 and ≤12 years of age at the time of informed consent/assent.
* Females of childbearing potential who are not pregnant and not nursing.
* Females of childbearing potential who agree to practice a clinically accepted method of contraception during the study and for at least 1 month prior to study dosing and 1 month following completion of the study. Acceptable contraceptive methods include abstinence, oral contraception, surgical sterilization (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), intrauterine device, or diaphragm in addition to spermicidal foam and condom on male partner, or systemic contraception (eg, levonorgestrel-releasing implant).
* Diagnosis of ADHD (any type: combined, predominately hyperactive impulsive type or predominately inattentive type) by a psychiatrist, psychologist, pediatrician, or licensed allied healthcare professional using the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) and confirmed by administration of a structured diagnostic interview using the Kiddie-Schedule for Affective Disorders and Schizophrenia for School Age Children-Present and Lifetime DSM-5 version (K-SADS-PL).
* Subjects who have received, or are receiving treatment with medication (amphetamine, methylphenidate, or non-stimulant) for ADHD must be willing to undergo a washout period of a minimum of 3 days or 5 half-lives (whichever is longer) prior to study drug administration. The washout period for prohibited concomitant medications will be at least 5 half-lives or 3 days, whichever is longer.
* If subjects are currently off treatment, this must be for any reason other than noncompliance, nonresponse, or intolerance to side effects.
* Ratings on the attention deficit/hyperactivity disorder-Rating Scale, version 5 (ADHD RS-5) when the subject is not receiving treatment for ADHD must be ≥90th percentile normative value for sex and age in at least 1 of the categories: total score, inattentive subscale, or hyperactive/impulse subscale.
* Dissatisfied with his or her current pharmacological therapy for treatment of ADHD or not currently receiving pharmacological therapy for ADHD for any reason other than nonresponse, noncompliance, or tolerability issues with stimulants. Newly diagnosed and treatment naïve subjects may be included at the discretion of the investigator.
* Must be functioning at an age-appropriate level intellectually as determined by an intelligence quotient (IQ) of ≥80 on a documented IQ assessment such as the Wechsler Abbreviated Scale of Intelligence II (WASI-II) vocabulary and matrix reasoning components, or the Kaufman Brief Intelligence Test, Second Edition (KBIT-2)
* Parent(s)/legal guardian(s) must have the ability to read and understand the language in which the informed consent is written and are mentally and physically competent to provide written informed consent for their child.
* Written or verbal assent from the subject (as applicable).
* Subject and parent(s)/legal guardian/caregiver are willing and able to comply with all the protocol requirements and parent(s)/legal guardian/caregiver must be able to provide transportation for the subject to and from the clinic visits.

Exclusion Criteria:

* Has a known allergy, intolerance, or hypersensitivity to methylphenidate.
* History of allergic reactions to tartrazine.
* Known nonresponder to methylphenidate treatment.
* Subject has received a monoamine oxidase inhibitor within 2 weeks before study treatment.
* Blood pressure and heart rate outside the 95th percentile for age and sex.
* Subject has a current or recent history (within the past 6 months) of drug abuse or dependence disorder; or someone in the subject's immediate family has a current or recent history (within the past 6 months) of drug abuse or dependence disorder; or someone living at the subject's home has a current or recent history (within the past 6 months) of drug abuse or dependence disorder; or subject has a positive urine drug screen for stimulant medication (other than currently prescribed stimulant for the treatment of ADHD) or drugs of abuse at the screening visit.
* Has abnormal thyroid function, glaucoma, Gilles de la Tourette's disorder, a history of seizures (except simple febrile seizures), or a tic disorder. Mild medication induced tics are not exclusionary.
* Primary and/or comorbid psychiatric diagnosis other than ADHD with the exception of simple phobias, motor skill disorders, communication disorders, learning disorders, and adjustment disorders so long as such disorder is judged not to interfere with study participation or the safety of the subject.
* Subjects with a family history (first-degree relatives) of sudden cardiac death require review and approval by the medical monitor for participation in the study.
* Subject has a history of disorders of the sensory organs, including deafness, blindness or the subject is severely or profoundly developmentally disabled.
* Any clinically significant abnormality or clinically significant abnormal laboratory test results found during screening or a positive test for hepatitis A, hepatitis B, hepatitis C, or HIV found during screening (subjects who have received a hepatitis A vaccine and test positive for hepatitis A may be included in the study, at the discretion of the investigator).
* Use of an investigational drug within 30 days (90 days for biologics) or participation in an investigational study within 30 days prior to dosing.
* Any reason which, in the opinion of the investigator, would prevent the subject from participating in the study.
* Clinically significant ECG abnormalities (including but not limited to Wolff Parkinson-White syndrome, supraventricular tachycardia, left ventricular hypertrophy, abnormal conduction defect, or other cardiac arrhythmia), or vital sign abnormalities (normal vital signs should be between 5th and 95th percentile for age) at screening.
* Known history of cardiovascular disorders including hypertension, angina, arterial occlusive disease, heart failure, hemodynamically significant congenital heart disease, cardiomyopathies, myocardial infarction, potentially life-threatening arrhythmias, and channelopathies (disorders caused by the dysfunction of ion channels).
* Clinically significant history of neurological, endocrinal (including thyrotoxicosis), pulmonary, hematological, immunologic, gastrointestinal, renal, hepatic or metabolic disease, or psychiatric illness other than ADHD.
* History of anxiety, tension, agitation, motor tics, Tourette's syndrome or a family history (first-degree relatives) of Tourette's syndrome.
* History of glaucoma.
* Has a positive serum pregnancy test (if applicable) at screening.
* Positive findings on the Columbia-Suicide Severity Rating Scale (C-SSRS) for suicidal ideation or behaviors at screening.
* Clinically significant illness or surgery within 4 weeks prior to dosing. Subjects who experience vomiting within 24 hours prior to clinic admission will be carefully evaluated for upcoming illness/disease.
* Hemoglobin <105 g/L or hematocrit <0.310 L/L at screening (subjects with abnormal hemoglobin and/or hematocrit levels deemed not clinically significant may be included in the study, at the discretion of the investigator).
* Subject has received anticonvulsants (eg, phenobarbital, phenytoin, primidone), coumarin anticoagulants, prescription pressor agents, pressor agents, guanethidine, tricyclic antidepressants (imipramine, desipramine, selective serotonin inhibitors) or herbal remedies within 30 days prior to the first dosing, or melatonin within 3 days prior to the first dosing.

Other protocol specific inclusion/exclusion criteria may apply.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - MCB Clinical Research Centers, LLC, Colorado Springs, Colorado
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Adaptive Clinical Research, Inc., Lauderhill, Florida
  - Accel Research Sites - Maitland Clinical Research Unit, Maitland, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Sisu BHR, LLC, Springfield, Massachusetts
  - Clinical Research of Southern Nevada, LLC, Las Vegas, Nevada
  - IPS Research Company, Oklahoma City, Oklahoma
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Family Psychiatry of the Woodlands, The Woodlands, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - Eastside Therapeutic Resource, Inc. dba Core Clinical Research, Everett, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject first visit: August 3, 2021; Last subject last visit: April 27, 2022. Thirteen investigative centers in the United States enrolled participants in the study.
  The study was terminated early due to administrative reasons unrelated to efficacy or safety.
Period: Overall Study
Arm/Group | Adhansia XR
Started | 103
Completed | 0
Not Completed | 103
Not completed — Study was Terminated by Sponsor | 103

BASELINE CHARACTERISTICS:
Arm/Group | Adhansia XR
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age for 1 subject was missing
  years
    number analyzed (Participants) | 102
    (all) | 9 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 37
  White | 60
  More than one race | 3
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Adverse Events as a Measure of Safety
Description: Adverse events (AEs) were documented and reported from the time the subject/parent(s)/legal guardian provided informed consent/assent up to 7 days after the last study drug administration. AEs that were ongoing at the subject's last study visit were followed until resolution or for 30 days after study drug administration.
Time Frame: Up to 9 months
Population: The safety analysis population is defined as all subjects who were administered at least 1 dose of study drug and had any safety information.
Measure: Number; unit: participants
Arm/Group | Adhansia XR
Number analyzed (Participants) | 103
participants
  Deaths | 0
  Serious Adverse Events | 2
  All Other Adverse Events in ≥ 5% of subjects | 39

ADVERSE EVENTS:
Time Frame: Documenting and reporting of AEs began when the subject/parent(s)/legal guardian provided informed consent/assent and continued up to 7 days after the last administration of study drug. Adverse events ongoing at the subject's last study visit must have been followed until resolution or for 30 days after study drug administration. Adverse events were collected for up to 9 months.
Arm/Group | Adhansia XR
All-Cause Mortality (participants affected / at risk) | 0/103
Serious Adverse Events (participants affected / at risk) | 2/103
Other Adverse Events (participants affected / at risk) | 39/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adhansia XR (N=103)
Suicidal Ideation (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adhansia XR (N=103)
Abdominal pain upper (Gastrointestinal disorders) | 10
Upper respiratory tract infection (Infections and infestations) | 8
Decreased appetite (Metabolism and nutrition disorders) | 17
Insomnia (Psychiatric disorders) | 18
Irritability (Psychiatric disorders) | 11

LIMITATIONS AND CAVEATS:
Study terminated early - only safety data collected until termination are presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT04987762/Prot_SAP_001.pdf